CLINICAL TRIAL: NCT01922284
Title: A Phase I Clinical Trial Investigating Immunisation Strategies Using DNA, MVA and CN54rgp140 Adjuvanted With GLA-AF to Maximise Antibody Responses
Brief Title: Investigating Immunisation Strategies of DNA, MVA and CN54rgp140 Adjuvanted With GLA-AF to Maximise Antibody Responses
Acronym: UKHVCSpoke003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRO2059; 2012-003277-26 (EudraCT Number)
Record Dates: First submitted 2013-07-10; First posted 2013-08-14 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2013-08

CONDITIONS: HIV
Keywords: HIV; Vaccine; Immunisation; DNA; Adverse events; MVA-C; GLA-AF; Antibody
MeSH Terms: interventions — DNA; GLA-AF adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Combination arm (Experimental): All participants will receive DNA vaccines at 0,4 and 8 weeks. These will be administered in 2 separate injections of 1ml (CN54ENV into the muscle of the upper right arm and ZM96GPN into the muscle of upper left arm). Participants in group 1 will receive 5 immunisations (DNA, MVA and CN54rgp140 in GLA-AF vaccines) at weeks 0, 4, 8 16 and 20.
  At weeks 16 and 20, individuals in group 1 will be given MVAC in a volume of 0.5mls into the upper left arm and also 100ug CN54rgp140 mixed with 5ug GLA-AF in a total volume of 0.4mls into the muscle of the upper right arm.
  Interventions: Biological: DNA; Biological: MVA-C; Biological: CN54rgp140; Biological: GLA-AF
- Group 2 - Non-combination arm (Active Comparator): All participants will receive DNA vaccines at 0,4 and 8 weeks. These will be administered in 2 separate injections of 1ml (CN54ENV into the muscle of the upper right arm and ZM96GPN into the muscle of upper left arm). Participants in group 2 will receive 7 immunisations (DNA, MVA and CN54rgp140 in GLA-AF vaccines) at weeks 0, 4, 8, 16, 20, 24 and 28.
  At weeks 16 & 20 group 2 will receive only 0.5mls of MVAC into the muscle of the upper left arm. At weeks 24 and 28 they will receive injections of 100ug CN54rgp140 mixed with 5ugGLAAF in a total volume of 0.4mls into the muscle of the upper right arm.
  Interventions: Biological: DNA; Biological: MVA-C; Biological: CN54rgp140; Biological: GLA-AF

INTERVENTIONS:
Biological: DNA — 8mg DNA: one plasmid encoding a gag-pol-nef polypeptide derived from the 96ZM651-8 clone and one plasmid encoding gp140 env derived from clade C 97CN54
Biological: MVA-C — 1.108 TCID50 MVA-C (nominal titre) expressing the gag-pol-nef and gp120 env proteins derived from clade C 97CN54
Biological: CN54rgp140 — 100ug CN54rgp140, a trimeric recombinant envelope protein derived from clade C 97CN54
Biological: GLA-AF — 5ug GLA-AF, an aqueous glucopyranosyl lipid A adjuvant

SUMMARY:
UKHVC Spoke 003 is a randomised Phase I, two centre study which will explore the impact of shortening a vaccination regimen using deoxyribonucleic acid (DNA) (CN54ENV and ZM96GPN), Modified Vaccinia Ankara - C (MVA-C) and CN54rgp140 adjuvanted with glucopyranosyl lipid A adjuvant - aqueous form (GLA-AF). The study population will be 40 healthy male and female volunteers 18 to 45 years old who are at low risk of HIV infection are to be recruited.

Study participants will be immunised with trial immunogens:

* 8mg DNA: one plasmid encoding a gag-pol-nef polypeptide derived from the 96ZM651-8 clone and one plasmid encoding gp140 env derived from clade C 97CN54
* 1.108 TCID50 MVA-C (nominal titre) expressing the gag-pol-nef and gp120 env proteins derived from clade-C 97CN54
* 100ug CN54rgp140, a trimeric recombinant envelope protein derived from clade C 97CN54
* 5ug GLA-AF, an aqueous glucopyranosyl lipid A adjuvant

All immunisations will be administered by the intramuscular route (IM). CN54gp140 and GLA will be mixed together before administration, and immunogens will be delivered in combination regimens

DETAILED DESCRIPTION:
This is a phase I study exploring the safety and potency of five HIV vaccines in healthy volunteers. The main aim is to see whether three of the five vaccines can be given together rather than one after the other, in five rather than seven sets of vaccinations and a course shortened by eight weeks. All volunteers will receive three injections of the first two vaccines (DNA plasmids) and half will be randomly assigned to receive two injections each of the second (MVA-C) and subsequent vaccines (CN54rgp140 mixed with GLA-AF) during the same visit or two injections of the MVA-C followed by two of CN54rgp140 mixed with GLA-AF.

The investigators are interested in ensuring that the vaccines are safe and also that the immune responses in the two groups of volunteers are similar. The three vaccines have all been shown to stimulate the immune response to specific parts of the HIV virus and none are infectious. The first vaccine consists of two DNA plasmids. When injected into muscle cells small parts of the HIV virus which are encoded by the DNA are produced and these are then recognised by the immune system. The second vaccine MVAC, is derived from vaccinia virus which has been modified so that it cannot divide. The virus (Modified Vaccinia Ankara (MVA)) actually expresses the same portions of HIV as the DNA and results in amplification of the responses seen. The third vaccine is a synthetically produced component of the HIV viral outer coat and it will be administered with an additive which has been shown to greatly enhance particular types of immune response which have recently been shown to play a role in protection against infection

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged between 18 and 45 years on the day of screening
2. Available for follow-up for the duration of the study (up to ~10 months from enrolment)
3. At low risk of HIV and willing to remain so for the duration of the study defined as:

   * no history of injecting drug use in the previous ten years
   * no gonorrhoea or syphilis in the last six months
   * no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months
   * no unprotected anal intercourse in the last six months, outside a relationship with a regular partner known to be HIV negative
   * no unprotected vaginal intercourse in the last six months outside a relationship with a regular known/presumed HIV negative partner
4. Willing to undergo an HIV test
5. Willing to undergo a genital infection screen if indicated by sexual history
6. If heterosexually active female, using an effective method of contraception with partner other than an IUCD/IUS (combined oral contraceptive pill; injectable or implanted contraceptive; consistent record with condoms if using these; physiological or anatomical sterility in self or partner) from 14 days prior to the first vaccination until 4 months after the last, and willing to undergo urine pregnancy tests prior to each vaccination
7. If heterosexually active male, using an effective method of contraception with their partner from the first day of vaccination until 4 months after the last vaccination
8. Agree to abstain from donating blood for three months after the end of their participation in the trial, or longer if necessary
9. Registered with a general practitioner (GP) for at least the past three months
10. Satisfactory response received from GP before randomisation
11. Willing and able to give written informed consent

Exclusion Criteria:

1. Pregnant or lactating
2. Presence of an IUCD (intrauterine contraceptive device)/IUS (intrauterine system)
3. Clinically relevant abnormality on history or examination including

   * history of grand-mal epilepsy, seizure disorder or any history of prior seizure
   * severe eczema
   * liver disease with inadequate hepatic function
   * any skin condition which may interfere with the trial assessment on the injection site
   * haematological, metabolic, gastrointestinal or cardio-pulmonary disorders
   * uncontrolled infection; toxic shock syndrome; autoimmune disease, immunodeficiency or use of immunosuppressives in preceding 3 months
4. Known hypersensitivity to any component of the vaccine formulations used in this trial, or have severe or multiple allergies to drugs or pharmaceutical agents
5. History of severe local or general reaction to vaccination defined as

   1. local: extensive, indurated redness and swelling involving the major circumference of the arm, not resolving within 72 hours
   2. general: fever >= 39.5°C within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
6. Receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of enrolment
7. Receipt of an experimental vaccine containing HIV antigens at any time in the past
8. Receipt of blood products or immunoglobin within 4 months of screening
9. Participation in another trial of a medicinal product, completed less than 30 days prior to enrolment
10. HIV 1 or 2 positive or indeterminate on screening
11. Positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
12. Grade 1 or above routine laboratory parameters. Hyperbilirubinaemia to be considered an exclusion criterion only when confirmed to be conjugated bilirubinaemia
13. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
14. Unlikely to comply with protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Magnitude of antibody response | Four weeks after final immunisation
  Magnitude (reciprocal mean endpoint titre and concentration) of systemic Immunoglobulin G (IgG) binding antibody responses to CN54rgp140 measured four weeks after the final immunisation.
Adverse Events | Every four weeks up to 32 weeks
  Grade 3 or above local solicited adverse event Grade 3 or above systemic clinical and laboratory solicited adverse event Any grade of adverse event that results in a clinical decision to discontinue further immunisations

SECONDARY OUTCOMES:
Magnitude of neutralising antibody (Nab) responses | Four weeks after the final immunisation
  Confirmation of specific investigations will be provided at a later date.
Magnitude of T-cell and B-cell responses | Four weeks after the final immunisation
  Confirmation of specific investigations will be provided at a later date.
Magnitude of mucosal IgG and IgA antibody responses | Four weeks after the final immunisation
  Confirmation of specific investigations will be provided at a later date.
Magnitude of antibody-dependent cell-mediated cytotoxicity or Antibody-dependent cell-mediated viral inhibition | From first immunisation
  Confirmation of specific investigations will be provided at a later date.
Magnitude of systemic Immunoglobulin A (IgA) binding antibody responses | Four weeks after the final immunisation
  Confirmation of specific investigations will be provided at a later date.

CONTACTS AND LOCATIONS:
Overall Officials: Sheena McCormack, MSc, FRCP, Principal Investigator — Senior Clinical Scientist
Locations (2):
- United Kingdom (2):
  - Surrey Clinical Research Centre, University of Surrey, Guildford, Surrey
  - Imperial College London, Greater London